CLINICAL TRIAL: NCT06486285
Title: Auditory-Cognitive Dual-Task Intervention for Older Adults With Hearing Loss: A Pilot Randomized Controlled Trial
Brief Title: Auditory-Cognitive Dual-Task Intervention for Older Adults With Hearing Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P0045159
Record Dates: First submitted 2024-06-18; First posted 2024-07-03 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2024-06

CONDITIONS: Age-related Hearing Loss; Cognitive Decline; Loneliness; Social Isolation
MeSH Terms: conditions — Presbycusis; Cognitive Dysfunction; Social Isolation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Auditory-cognitive dual-task training (ACDT) (Experimental): The new auditory-cognitive dual-task training (ACDT) is a 12-week program (5 times/week, 60 minutes per day). Auditory training (i.e., speech-in-noise training, rapid speech training and competing speaking training) will be incorporated with cognitive exercises involving the domains of executive function, perceptual-motor ability, memory, and complex attention.
  Interventions: Behavioral: Auditory-cognitive dual-task training (ACDT)
- Control (No Intervention): no specific treatment. This is a "wait list" group, participants can choose either the Auditory-cognitive dual-task training or the cognitive training after 12 weeks.

INTERVENTIONS:
Behavioral: Auditory-cognitive dual-task training (ACDT) — The components of auditory training are designed based on an auditory training and aural rehabilitation program LACETM (Listening & Communication Enhancement) developed by our study team member. The cognitive training was developed and tested feasible and valid in our study team's previous dual-task Zumba cognitive training.
  Arms: Auditory-cognitive dual-task training (ACDT)

SUMMARY:
Background: Age-related hearing loss (ARHL) is a common and irreversible condition that has been recently associated with cognitive decline and dementia. Hence, if ARHL is treated earlier, the risk of dementia might decrease. However, in China, only 0.8% of older adults with hearing loss wore hearing aids, and over two-thirds (67.5%) of older adults with ARHL in Hong Kong had either been formally diagnosed or treated. There is also limited information on the feasibility and efficacy of hearing loss interventions for older people in Hong Kong. It is important to develop hearing loss interventions that have the potential to improve cognitive functions among older people.

Aims: This study aims to assess the feasibility and acceptability of a new auditory-cognitive dual-task intervention (ACDT) for community-dwelling older adults with hearing loss, and to examine the preliminary efficacy of ACDT on their cognitive function.

Study design and Methods: This is mixed-model design, using a 2-arm, parallel-group, single-blinded, pilot randomized controlled trial (pilot RCT). A total of 60 community-dwelling older adults in Hong Kong who have mild to moderate hearing loss and normal cognitive performance will be recruited. Participants will be randomly assigned to the auditory-cognitive dual-task intervention group (ACDTG), and control group with no specific intervention (a "wait list" group) (CG). Each ACDTG participant will receive the intervention for 12 weeks (5 days x 60-min sessions per day). All participants in all groups will be assessed for cognitive function (primary outcome), social isolation, and loneliness, and hearing at baseline (T0), and after the intervention (T1). Post-intervention interviews will be conducted to obtain perspectives of participants in the ACDTG on the feasibility and acceptability of the ACDT intervention.

Data analysis: Participant characteristics and outcome variables will be analysed through descriptive statistics. Differences in cognition score and other outcomes across time points among the participant groups will be measured by Generalized Estimating Equations (GEE). The statistical software package IBM SPSS version 26.0 will be used. Content analysis will used to analyse the post-intervention interviews.

Expected results: ACDT will be feasible for implementation and acceptable for community-dwelling older adults with hearing loss. While ACDT will not be able to improve underlying hearing in ARHL, it will be more effective on improving participants' cognitive function, social engagement and loneliness, and ability in information processing, interpretation and communication, than CG.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 and above living in the community;
* have mild to moderate hearing loss with a pure-tone average (PTA) between 25 and 60 dB in both ears (average hearing threshold at 0.5, 1, 2, and 4 kHz measuring by audiometer with headphones in a quite listening environment, no hearing aid use within the past 6 months;
* with normal cognitive performance (MoCA score ≥26); and
* are willing to and capable of providing informed consent and complying with study procedures.

Exclusion Criteria:

* have a history of psychosis, mania, bipolar disorder, substance use disorder or have current suicidal ideation;
* with severe or unstable medical illness, significant retrocochlear pathology or organic lesion responsible for hearing loss;
* a diagnosis of probable Alzheimer's disease, vascular dementia, FTD, or Parkinson's Disease; and
* taking medications such as antidepressants, sedatives, or antiepileptics that may affect cognition.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Global cognition | will be assessed at baseline (T0), and Week 12 (immediately after the intervention) (T1)
  Global cognition will be measured by the Hong Kong-Montreal Cognitive Assessment (HK-MoCA). MoCA measures multiple cognitive domains, including attention, orientation, concentration, language, memory, executive functions and visuo-spatial skills. MoCA ≥26 is considered as normal, while 22-26 refers to mild cognitive impairment.

SECONDARY OUTCOMES:
Learning and memory | will be assessed at baseline (T0), and Week 12 (immediately after the intervention) (T1)
  The Chinese Auditory Verbal Learning Test will be used.
Hearing | will be assessed at baseline (T0), and Week 12 (immediately after the intervention) (T1)
  will be measured by an audiometer with sound level meter (to measure ambient noise).
Social isolation | will be assessed at baseline (T0), and Week 12 (immediately after the intervention) (T1)
  will be measured by validated abbreviated 6-item Chinese version of the Lubben Social Network Scale (LSNS), which was developed specifically for use among older adults and shown to be both reliable and valid.The total score is calculated by finding the sum of the all items. For the LSNS-R, the score ranges between 0 and 60, with a higher score indicating more social engagement. For the LSNS-6, the score ranges between 0 and 30, with a higher score indicating more social engagement.
Loneliness | will be assessed at baseline (T0), and Week 12 (immediately after the intervention) (T1)
  will be measured by the 6-item De Jong Gierveld loneliness scale (Chinese version). The total score of the scale ranges from zero to six, with higher scores indicating greater feelings of loneliness. A cut-off score of two or more was used to indicate the presence of loneliness, as recommended by van Tilburg and De Jong Gierveld
Hearing | will be assessed at baseline (T0), and Week 12 (immediately after the intervention) (T1)
  Chinese version of the Hearing Handicap Inventory for the Elderly and the five-point Communication Scale for Older Adults will be utilized. The questionnaire consists of 10 items-five social/situational items and five emotional response items-with a total score range of 0-40. A "YES" response receives four points, a "NO" response receives zero points, and a "SOMETIMES" response receives two points. The HHIE-S total scores were used to classify the results into three categories: 0 to 8 (no self-perceived hearing handicap), 10-24 (mild to moderate handicap), and 26-40 (severe handicap). According to the American Speech-Language-Hearing Association's proposed recommendations, a total HHIE-S score of 8 indicates the presence of a hearing handicap
Attention or working memory | will be assessed at baseline (T0), and Week 12 (immediately after the intervention) (T1)
  will be measured by the digit span (forward and backward) and visual span (forward and backward) methods
Information processing speed | will be assessed at baseline (T0), and Week 12 (immediately after the intervention) (T1)
  will be assessed by the performance on the Chinese Trail Making Test Part A
Executive function | will be assessed at baseline (T0), and Week 12 (immediately after the intervention) (T1)
  Will be assessed by the Chinese Trail Making Test Part B
Verbal fluency | will be assessed at baseline (T0), and Week 12 (immediately after the intervention) (T1)
  will be assessed by the category verbal fluency tests (animal, fruit, and vegetable)
Motor skills | will be assessed at baseline (T0), and Week 12 (immediately after the intervention) (T1)
  will be evaluated by the grooved pegboard for both dominant hand and nondominant hand

CONTACTS AND LOCATIONS:
Overall Officials: Ivy Zhao, Dr, Principal Investigator — School of Nursing, the Hong Kong Polytechnic University
Locations (1):
- PolyU, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Individual deidentified participant data (including data dictionaries) will be shared. The investigators will publish research findings in peer reviewed and international official journals without Individual identifiable participant information according to the ethical requirement. Individual deidentified participant dataset can be shared per request and approved by the research core team.